CLINICAL TRIAL: NCT01564836
Title: A Multi-center Study of the Discontinuation of Imatinib in Adult Patients With Ph+ CML in CP Who Have a Complete Molecular Response to Imatinib
Brief Title: Discontinuation Study of Imatinib in Adult CP CML Patients Who Have a Complete Molecular Response to Imatinib
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Dong-Wook Kim, Professor, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC10ENME0465
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Myeloid Leukemia; Imatinib; Complete Molecular Response
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib treatment discontinuing (Experimental)
  Interventions: Behavioral: Imatinib treatment discontinuing

INTERVENTIONS:
Behavioral: Imatinib treatment discontinuing — Ph+ CP CML patients who were treated with IM for more than 3 years in sustained MR4.5 or undetectable transcript for at least 2 years are enrolled

SUMMARY:
This prospective study is performed to identify safer and more concrete indicators of successful discontinuation and explore contributing factors for sustained undetectable transcript

DETAILED DESCRIPTION:
Imatinib (IM) treatment has been the standard of care for chronic phase (CP) chronic myeloid leukemia (CML) and approximately 50% of CP CML patients who received IM treatment achieve complete molecular response (CMR) at 6-7 years.(Hochhaus A et al. Leukemia 2009;23:1054-1061, Hughes et al. Blood 2008;112:334) The recent data from a study aimed to assess whether IM can be discontinued in patients with a CMR lasting at least 2 years showed the probability of persistent CMR at 12 months was 41%, and suggested IM can be safely discontinued, at least in some patients with sustained CMR. (Mahon et al. Lancet Oncol 2010;11:1029-1035) However, to define whether discontinuation of IM treatment can be safely employed, further validation and much longer follow-up are needed.

Aims This prospective study is performed to identify safer and more concrete indicators of successful discontinuation and explore contributing factors for sustained undetectable transcript.

Primary Objective:

* To evaluate the probability of persistent undetectable molecular residual disease (UMRD) and MR4.5 at 12 months after discontinuation
* To measure the duration of persistent UMRD and MR4.5 after discontinuation
* To identify contributing factors for sustained undetectable transcript

Secondary Objective:

* To evaluate the probability of major molecular response (MMR) loss
* To evaluate the time taken to lose MMR at 12 months after discontinuation
* In patients with loss of MMR, the probability of re-achieving MMR/MR4.5
* To measure the time taken to re-achieve MMR/MR4.5 after IM resumption
* To identify contributing factors for sustained re-achieve MMR/MR4.5

Trial Design This is a prospective, multicenter, non-randomised IM discontinuation study.

Response Evaluation After discontinuation, molecular response was monitored using RQ-PCR assay every month up to 6 month follow-up, every 2 months up to 12 month follow-up, and every 3 months thereafter. The loss of MMR, MR4.5, and UMRD were defined on 2 consecutive assessments.

If loss of MMR occurred, IM treatment was re-introduced. Written informed consents were obtained for all patients

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years-old) Ph+ CP CML patients who were treated with IM for more than 3 years in sustained MR4.5 or undetectable transcript for at least 2 years are enrolled. MR4.5 or undetectable transcript must be sustained by 2 consecutive RQ-PCR assay within 6 months

Exclusion Criteria:

* Patients were diagnosed with AP or BP CML
* Ph+ ALL
* Received cytotoxic chemotherapy or any other TKIs except imatinib
* Any evidence of on-going graft versus-host disease (GVHD)
* Relapsed patients after allogeneic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Probability of persistent undetectable molecular residual disease (UMRD) and MR4.5 | 12 months
  Our primary objectives were to evaluate the probability of persistent undetectable molecular residual disease (UMRD) and MR4.5 at 12 months after discontinuation, to measure the duration of persistent UMRD and MR4.5 after discontinuation, and to identify contributing factors for sustained undetectable transcript.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee SE, Choi SY, Song HY, Kim SH, Choi MY, Park JS, Kim HJ, Kim SH, Zang DY, Oh S, Kim H, Do YR, Kwak JY, Kim JA, Kim DY, Mun YC, Lee WS, Chang MH, Park J, Kwon JH, Kim DW. Imatinib withdrawal syndrome and longer duration of imatinib have a close association with a lower molecular relapse after treatment discontinuation: the KID study. Haematologica. 2016 Jun;101(6):717-23. doi: 10.3324/haematol.2015.139899. Epub 2016 Feb 17. PMID 26888022